CLINICAL TRIAL: NCT02755077
Title: Effect of Head Rotation on Efficiency of Face Mask Ventilation in Anesthetized Apneic Adults: A Prospective Randomized Crossover Study
Brief Title: Effect of Head Rotation on Efficiency of Face Mask Ventilation in Anesthetized Apneic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeremi R Mountjoy, M.D., Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2013P002571
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Anesthesia
Keywords: Anesthesia induction; Airway; Mask ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mask ventilation in rotated head position (Experimental): Patient's head will be axially rotated 45 degrees to the right
  Interventions: Procedure: Head rotation during mask ventilation
- Mask ventilation in neutral head position (No Intervention)

INTERVENTIONS:
Procedure: Head rotation during mask ventilation — Patient's head position is axially rotated 45 degrees to the right.
  Arms: Mask ventilation in rotated head position

SUMMARY:
Upper airway obstruction commonly occurs after induction of general anesthesia. The aim of this study is to determine if head rotation improves the efficiency of mask ventilation of anesthetized apneic adults.

DETAILED DESCRIPTION:
When apnea is achieved after induction, face mask ventilation is started in either a neutral head position or a head position axially rotated 45 degrees to the right. Mask ventilation will be carried out for 1 minute (Step 1) with pressure control ventilation of an anesthesia machine at peak inspiratory pressure 15 cmH2O, 10 breaths per minute, inspiration time to expiration time ratio 1:2 and no positive end-expiratory pressure. Then, mask ventilation will continue but head position will be crossed over (Step 2) and Step 1 will be repeated (Step 3). Expiratory tidal volume (VTE) will be measured by using respiratory inductive plethysmograph.

ELIGIBILITY:
Inclusion Criteria:

* Patients with body mass index in the range of 18.5 to 35.0 kg/m2, who meet American society of anesthesiologists physical status classification I to III and require general anesthesia with tracheal intubation.

Exclusion Criteria:

* Patients with limited head rotation/extension, gastro-esophageal reflux or a full stomach, known sleep apnea in continuous positive airway pressure therapy and any anticipated difficult airway likely requiring awake intubation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in averaged expiratory tidal volume measured by Respiratory monitor | 1, 2 and 3 min after the initiation of mask ventilation
  Change in tidal volume between data of 2 min and average data from 1 and 3 min

CONTACTS AND LOCATIONS:
Overall Officials: Jeremi R Mountjoy, M.D., Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Isono S, Tanaka A, Nishino T. Lateral position decreases collapsibility of the passive pharynx in patients with obstructive sleep apnea. Anesthesiology. 2002 Oct;97(4):780-5. doi: 10.1097/00000542-200210000-00006. PMID 12357140
- [Background] Walsh JH, Maddison KJ, Platt PR, Hillman DR, Eastwood PR. Influence of head extension, flexion, and rotation on collapsibility of the passive upper airway. Sleep. 2008 Oct;31(10):1440-7. PMID 18853942
- [Derived] Itagaki T, Oto J, Burns SM, Jiang Y, Kacmarek RM, Mountjoy JR. The effect of head rotation on efficiency of face mask ventilation in anaesthetised apnoeic adults: A randomised, crossover study. Eur J Anaesthesiol. 2017 Jul;34(7):432-440. doi: 10.1097/EJA.0000000000000582. PMID 28009638